CLINICAL TRIAL: NCT06482268
Title: An Investigator-initiated Clinical Trial of Safety and Efficacy of Transplantation of Human Induced Pluripotent Stem Cell-derived Dopaminergic Progenitors (CT1-DAP001) for Parkinson's Disease (Phase I/II)
Brief Title: Transplantation of Human iPS Cell-derived Dopaminergic Progenitors (CT1-DAP001) for Parkinson's Disease (Phase I/II)
Acronym: CT1-DAP001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry); Kyoto University (Other); Sumitomo Pharma Co., Ltd. (Industry); CiRA Foundation (Unknown)
Responsible Party: Principal Investigator, Joseph Ciacci, Program Director/Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 808955
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: PD - Parkinson's Disease
Keywords: Parkinson's Disease; Ataxia; Dopaminergic; Dyskinesia; PD; Neurodegenerative Disease; Brain Disease; CNS; Movement Disorder; Central Nervous System Disease; FDOPA; MRI; Corpus striatum
MeSH Terms: conditions — Parkinson Disease; Ataxia; Dyskinesias; Neurodegenerative Diseases; Brain Diseases; Movement Disorders; Central Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a single-center, open-label, uncontrolled study to evaluate the safety of transplantation of CT1-DAP001 as the primary objective, and as a secondary objective, to evaluate efficacy. Seven (7) subjects with PD will be followed up for 24 months after transplantation of approximately 4.2-5.4 × 106 dopaminergic progenitors per side into the bilateral putamen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-center, open-label, uncontrolled (Other): To evaluate the safety and efficacy of transplantation of human induced pluripotent stem cell-derived dopaminergic progenitors, CT1-DAP001, into the corpus striatum in patients with Parkinson's disease
  Interventions: Combination Product: Human induced pluripotent stem cell-derived dopaminergic progenitors (CT1-DAP001)

INTERVENTIONS:
Combination Product: Human induced pluripotent stem cell-derived dopaminergic progenitors (CT1-DAP001) — Investigational PET agents will be synthesized at UCSD and administered to subjects according to the local institutional guidelines. IND applications for these agents are linked with the IND application for the study product, CT1-DAP001. The IND applications for the PET radiopharmaceuticals contains the manufacturing method, specifications, quality testing, clinical usage, and safety and efficacy information for individual PET agents.
  Investigational Cell Injector Suniviion needle: The investigational instrument will be used to administer dopaminergic progenitors into the putamen. After aspirating cells, the instrument will be attached to a Leksell stereotactic frame to administer the cells into the brain.
  Other Names: Investigational imaging - FDOPA & FEPPA; Investigational device - Sunovion needle

SUMMARY:
To evaluate the safety and efficacy of transplantation of human induced pluripotent stem cell-derived dopaminergic progenitors, CT1-DAP001, into the corpus striatum in patients with Parkinson's disease

DETAILED DESCRIPTION:
Single-center, open-label, uncontrolled. The primary objective of this study is to evaluate the safety of CT1-DAP001 in subjects with Parkinson's disease by determining the incidence and severity of adverse events, especially graft expansion, after transplantation into the corpus striatum. Other objectives are to evaluate the efficacy of CT1-DAP001 through the assessment of Parkinson's disease symptoms and clinical severity or progression.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a diagnosis of PD (clinically established or clinically probable) in accordance with the MDS Clinical Diagnostic Criteria for Parkinson's Disease (2015).
2. The subject has an inadequate response to drug treatments.
3. The subject is ≥ 40 years and ≤ 75 years of age at the time of informed consent.
4. The subject has had PD for at least 5 years.
5. The subject has both ON and OFF (as demonstrated by the MDS-UPDRS Part III and a symptom diary).
6. The subject does not have a debilitating dyskinesia score greater than or equal to 3 on the MDS-UPDRS.
7. The subject is in stage 2 or higher on the Hoehn and Yahr scale at OFF time.
8. The subject is in stage 3 or lower on the Hoehn and Yahr scale at ON time.
9. The subject has an L-dopa response of 30% or more without influence of antiparkinsonian drugs.
10. The subject has the following organ functions as determined by laboratory tests at Screening visit:

    1. Neutrophil count ≥ 2,000/μL
    2. Platelet count ≥ 5.0 × 104/μL
    3. AST, ALT ≤ 3.0 × upper limit of normal
    4. Total bilirubin ≤ 1.5 × upper limit of normal
    5. eGFR ≥ 60 mL/min/1.73 m2 (As part of Creatinine testing, an estimated glomerular filtration rate (mL/min/1.73 m2)will be calculated based on the CKD-EPI 2021 equation)
11. The subject is willing to avoid pregnancy using abstinence, highly effective means of birth control, surgical sterility, or menopause.
12. The subject is willing to comply with the protocol-required assessments.
13. The subject provides written informed consent to participate in the study. If the subject cannot sign due to physical constraints, verbal consent may be provided with signature of a Legally Authorized Representative.

Exclusion Criteria:

1. The subject has an abnormal brain MRI suggestive of brain pathology other than Parkinson's disease.
2. Atypical parkinsonism (Parkinsonism-Plus syndrome, secondary parkinsonism, hereditary parkinsonism).
3. The subject has clinical indication or diagnosis of abnormal immune function.
4. The subject has been diagnosed with a major neurocognitive disorder such as dementia, or is high risk for this.
5. The subject has bleeding tendency or abnormal coagulation function as evidenced by platelets <50 or PT/PTT > 1.5x normal.
6. The subject is HBs antigen-positive, or HBs antibody- or HBc antibody-positive with evidence of HBV-DNA.
7. The subject is anti-HIV antibody positive.
8. The subject is anti-HTLV-1 antibody-positive.
9. The subject has active infection such as hepatitis C or syphilis (STS/TPHA).
10. The subject has hypersensitivity or contraindication to tacrolimus, concomitant drugs (e.g., levodopa, carbidopa, MRI contrast), and/or their components.
11. Contraindications to general anesthesia as evaluated by subject matter experts.
12. The subject has a serious allergy to a component (e.g., gentamicin, component of bovine origin, or component of porcine origin) used in the preparation of the study product.
13. The subject has any of the following conditions/diseases concurrently:

    1. Malignant neoplasm
    2. Epilepsy
    3. Psychiatric disease (e.g., uncontrolled anxiety or depression, bipolar disorder, schizophrenia)
    4. Diabetes mellitus with poorly controlled blood glucose (glycosylated hemoglobin > 9.0%, or fasting plasma glucose (FPG) ≥ 200 mg/dL (11.1 mmol/L).
    5. Other serious concurrent diseases (e.g., cerebrovascular disorder, heart disease, chronic respiratory disease, inadequately controlled hypertension) as determined by the investigator.
14. The subject has a history of any of the following:

    1. Prior malignancy < 5 years prior to Screening. Patients who had prior malignancies within 5 years and in complete remission with expected survival of more than 5 years are not excluded
    2. Epilepsy
    3. Cerebral hemorrhage or stroke
    4. Psychiatric disease (e.g., uncontrolled anxiety or depression, bipolar disorder, schizophrenia)
    5. Congenital long QT syndrome
    6. Pallidotomy, thalamotomy, or Deep Brain Stimulation
15. The subject is pregnant or lactating or does not agree to avoid pregnancy throughout the study.
16. The subject has undergone transplantation of human iPSC-derived dopaminergic progenitors.
17. The subject, in the opinion of the investigator or sub investigator, is not appropriate to conduct the study safely.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
ACCEPTABILITY | 24 months
  Assessed by presence or absence of graft expansion (> 3 cm3) in the brain at 24 months after transplantation
SAFETY | 24 months
  Incidence and severity of treatment emergent adverse events assessed by graft expansion and size in the corpus striatum.

SECONDARY OUTCOMES:
QUALITY OF LIFE | 24 months
  Assessed by dyskinesia score, measured as the change in dyskinesia score from Baseline to each post-transplantation time point.
ACCURACY | 24 months
  Assessed by FDOPA (MRI) of tissue expansion The expansion on MRI will be assessed at each time point of measurement
  * day before transplantation,
  * immediately after transplantation,
  * day after transplantation,
  * 4 weeks, 12 weeks, 6 months, 18 months, (if clinically indicated)
  * 12 months, 24 months after transplantation
MDS-UPDRS Part III totalscore (at OFF time) | 24 months
  This endpoint is defined as the change in UPDRS Part III score at OFF time from Baseline to each post-transplantation time point. The efficacy will be assessed based on MDS-UPDRS Part III total score at OFF time at 24 months after cell transplantation.
  1. Excellent response defined as a decrease of ≥ 5
  2. Good response defined as a decrease of 0 to 4
MDS-UPDRS Part III totalscore (at ON time) | 24 months
  This endpoint is defined as the change in UPDRS Part III score at ON time from Baseline to each post-transplantation time point.
Average daily ON duration (with or without dyskinesia) and OFF duration | 24 months
  This endpoint is defined as the change in daily ON duration (with or without dyskinesia) or OFF duration from Baseline to each post-transplantation time point.
L-dopa equivalent dose | 24 months
  This endpoint is defined as the change in L-dopa equivalent dose from Baseline to 4 weeks, 12 weeks, 6 months, 12 months, 18 months, or 24 months after transplantation.
  Formula to convert to the L-dopa dose:
  L-dopa 100 mg = pramipexole salt 1 mg = ropinirole 5 mg = rotigotine 7.5 mg = bromocriptine 10 mg = pergolide 1 mg = cabergoline 1.5 mg = selegiline 10 mg = amantadine 100 mg = apomorphine 10 mg

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ciacci, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- See also: Parkinson's disease and related disorders (3) Parkinson's disease — http://www.nanbyou.or.jp/entry/314
- See also: Pre-clinical study of induced pluripotent stem cell- derived dopaminergic progenitor cells for Parkinson's Disease — http://www.neurology-jp.org/guidelinem/parkinson.html